CLINICAL TRIAL: NCT01195896
Title: A Prospective, Open, Non-controlled Clinical Investigation to Evaluate a New Negative Pressure Wound Therapy (NPWT) System to be Used in the Treatment of Acute Non-infected Wounds and Post Surgical Infected Wounds.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Molnlycke Health Care AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NPWT 02
Record Dates: First submitted 2010-09-03; First posted 2010-09-06 (Estimated); Last update posted 2012-01-16 (Estimated); Status verified 2012-01

CONDITIONS: Acute Non Infected Wounds; Non Infected Post Surgical Wounds

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: New NPWT system — According clinical routine (Instruction for Use)

SUMMARY:
The investigation is designed as a prospective, open, non-controlled clinical investigation.

DETAILED DESCRIPTION:
Wounds to be treated under this protocol should be acute non-infected wounds or post surgical infected wounds in hospitalized subjects. One ulcer per subject will be treated for a maximum duration of 3 weeks. All subjects will receive continuous negative pressure treatment with the new NPWT system with a pressure level of -120 mmHg or according to clinicians' instruction based on the indication.

10-15 subjects at two sites will be enrolled provided that they fulfil all the inclusion criteria and none of the exclusion criteria and who have signed and dated a written informed consent.

The subjects will be consecutively allocated to a specific subject identification code. The primary variable wound healing and granulation tissue formation will be assessed by digital planimeter, digital photography and visual estimation.

Subject pain will be measured by using the Visual Analogue Scale, VAS. Subject and investigator convenience will be assessed by convenience surveys. Diagnosis and treatment of wound infections according to clinical routine.

ELIGIBILITY:
Inclusion Criteria:

1. Acute non infected wound or infected post surgical wound suitable for Negative Pressure Wound Therapy according to the investigator's judgment
2. 3 cm2 ≤ Wound size ≤ 300 cm2
3. Male or female ≥18 years
4. Signed Informed Consent Form

Exclusion Criteria:

1. Need for frequent dressing changes, i.e.<48 hours between the changes
2. Dry wounds
3. Malignancy in the wound and/or wound margin
4. Untreated osteomyelitis
5. Untreated infection waiting for other intervention
6. Unexplored fistulas
7. > 10% necrotic tissue with eschar present after debridement
8. High risk for bleeding complications (including subject treated with anticoagulants that are associated with high risk for bleeding complications)
9. Exposed blood vessels, organs or nerves
10. Current or within 3 months treatment with chemotherapy or irradiation
11. Known hypersensitivity to the dressing material
12. Expected technically impossible to seal the film to achieve a vacuum treatment
13. Expected non compliance with the Clinical Investigation Plan
14. Pregnancy
15. Subjects previously included in this investigation
16. Subjects included in other ongoing clinical investigation at present or during the past 30 days
17. Target ulcer previously not successfully treated with NPWT within 48 hours from NPWT start
18. Subject unable to understand written patient information due to medical condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2010-09; Primary Completion 2011-08 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Granulation tissue formation | maximum 3 weeks
  To assess the wound healing and granulation tissue formation when using the NPWT system

SECONDARY OUTCOMES:
Handling of NPWT system | maximum 3 weeks
  To investigate the pain level at dressing removal To visually check exudate removal To investigate the ease of use for the subject and care giver when using the NPWT system

CONTACTS AND LOCATIONS:
Overall Officials: Mark Bischoff, Prof. Dr. med, Principal Investigator — Ulm University Hospital
Locations (1):
- Ulm University Hospital, Ulm, Germany